CLINICAL TRIAL: NCT01994161
Title: Clinical Registration Trial of Intracranial Stenting for Patients With Symptomatic Intracranial Artery Stenosis:A Prospective Multi-center, Registry Trial
Brief Title: Clinical Registration Trial of Intracranial Stenting for Patients With Symptomatic Intracranial Artery Stenosis(CRTICAS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XW125-S003
Record Dates: First submitted 2013-10-14; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; intracranial stenting; vascular risk factor management
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intracranial stenting group: all the participants in this group will be performed with intracranial stenting
  Interventions: Procedure: intracranial stenting

INTERVENTIONS:
Procedure: intracranial stenting — all the participants in this group will be performed with intracranial stenting
  --------------------------------------------------------------------------------

SUMMARY:
This trial is an prospective, government-funded registration study that will observe the safety and effectiveness of intracranial stenting for preventing stroke during a mean follow-up of 12 months in patients with symptomatic stenosis of a major intracranial artery (MCA, carotid, vertebral, basilar). This trial will be launched by Xuanwu Hospital, Capital University of Medical Science, with 20 collaborators participating. Enrollment will begin in 2013, and it aims to have a sample size of 840 subjects in 2 years. The trial is scheduled to complete in 2015.

As we know, SAMMPRIS is flawed with defect in design, heterogeneity in experience and credentials of operators and high rate of complication; Whether the interventional therapy for symtomatic intracranial artery stenosis is effective or not remained resolved. This trial has been modified based on SAMMPRIS in order to acquire the data for China: Technique, experience, and credential of the operators are closely related with perioperative complications in PTAS. The investigators select 50 large-scale medical centers for participation on the basis of geographical distribution. All the participants are ranked as top in China. They have the most experienced surgeons or interventionist in China, and are fully qualified for this trial. This will guarantee the success and safety of technique, maintain the continuity of operator's experience, and make the complication rate as low as possible.

DETAILED DESCRIPTION:
Title:Clinical Registration Trial of Intracranial Stenting for Patients With Symptomatic Intracranial Artery Stenosis:A Prospective Multi-center, Registry Trial

Design of trial:

This trial is an prospective, government-funded registration study that will observe the safety and effectiveness of intracranial stenting for preventing stroke during a mean follow-up of 3 years in patients with symptomatic stenosis of a major intracranial artery (MCA, carotid, vertebral, basilar). This trial was launched by Xuanwu Hospital, Capital University of Medical Science, with 40 collaborators participating. Enrollment will begin in 2013, and it aims to have a sample size of 840 subjects in 2 years. The trial is scheduled to complete in 2015.

Details:

SAMMPRIS (Stenting vs. Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis) hasn't received the expected results; But, it does not mean that angioplasty with stent on intracranial treatment come to a full stop. On the contrary, a discrepancy on reported data between multi-centre RCT and most single center studies urges us for thorough investigation in future.

As we know, SAMMPRIS is flawed with defect in design, heterogeneity in experience and credentials of operators and high rate of complication; Some questions about SAMMPRIS have been raised, and remained unresolved.

This trial has been modified based on SAMMPRIS in order to acquire the data for China: Technique, experience, and credential of the operators are closely related with perioperative complications in PTAS. The investigators select 40 large-scale medical centers for participation on the basis of geographical distribution. All the participants are ranked as top in China. They have the most experienced surgeons or interventionist in China, and are fully qualified for this trial. This will guarantee the success and safety of technique, maintain the continuity of operator's experience, and make the complication rate as low as possible.

SAMMPRIS was stopped ahead of schedule due to the safety concern. More than half of the PTAS patients were lost for follow-up at 1 year, and the remaining were followed up with a mean duration less than 1 year. It leaves the question of long-time follow-up data open. Base on SAMMPRIS, the investigators' trial will conduct a systematic follow-up system. Upon recruitment, all the patients' neurological and imaging examination will be determined at baseline, 1 week, 1 month, 6 months , 12 months after surgery, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic status: as evidenced by TIA or non-severe stroke within the past 12 months attributed to 70% to 99% stenosis of a major intracranial artery (carotid artery, MCA stem [M1], vertebral artery, or basilar artery).
* Degree of stenosis: 70%-99%; (Stenosis must be confirmed by catheter angiography for enrollment in the trial,WASID method)
* Age:30-80 years;
* No fresh infarctions identified on MRI (indicated as high signals on DWI series) upon enrollment
* No massive cerebral infarction (>1/2 MCA territory), intracranial hemorrhage, epidural or sub-dural hemorrhage, and intracranial brain tumor on CT or MRI scan
* mRS scale score of <=2
* Target vessel reference diameter must be measure d to be 2.00 mm to 4.50 mm; target area of stenosis is <=14 mm in length
* Patient is willing and able to return for all follow-up visits required by the protocol
* Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.

Exclusion Criteria:

* Untoward reaction to anesthesia.
* Any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe.
* Tandem extracranial or intracranial stenosis that is proximal or distal to the target intracranial lesion
* Previous treatment of target lesion with a stent, angioplasty, or other mechanical device.
* Any aneurysm proximal to or distal to stenotic intracranial artery. Intracranial tumor (except meningioma) or any intracranial vascular malformation
* Computed tomographic or angiographic evidence of severe calcification at target lesion
* Stroke of sufficient size (>5cm on CT or MRI) to place patient at risk of hemorrhagic conversion during the procedure.Hemorrhagic transformation of an ischemic stroke within the past 15 days.
* Previous spontaneous intracerebral (parenchymal) or other intracranial (subarachnoid, subdural, or epidural) hemorrhage within 30 days
* Untreated chronic subdural hematoma >5 mm in thickness
* Intracranial arterial stenosis related to arterial dissection, moya-moya disease or any known vasculitic disease;
* MI within previous 30 days
* Any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation
* Intolerance or allergic reaction to any of the study medications, including aspirin, clopidogrel, heparin, nitinol, and local or general anaesthesia History of life-threatening allergy to contrast dye. If not life-threatening and can be effectively pretreated, patient can be enrolled at physicians discretion
* Recent GI bleed that would interfere with antiplatelet therapy. Active bleeding diathesis or coagulopathy; active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets count <125,000, hematocrit <30, Hgb <10 g/dl, uncorrected INR >1.5, bleeding time >1 minute beyond upper limit normal, or heparin-associated thrombocytopenia that increases the risk of bleeding, uncontrolled severe hypertension (systolic BP>180 mm hg or diastolic BP>115 mm hg), severe liver impairment (AST or ALT >3 times normal, cirrhosis), creatinine >265.2μmol/l (unless on dialysis)
* Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 90 days after enrollment
* Severe dementia or psychiatric problem that prevents the patient from following an outpatient program reliably
* Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This trial is an prospective, government-funded registration study that will observe the safety and effectiveness of intracranial stenting for preventing stroke during a mean follow-up of 3 years in patients with symptomatic stenosis of a major intracranial artery (MCA, carotid, vertebral, basilar). This trial was launched by Xuanwu Hospital, Capital University of Medical Science, with 20 collaborators participating. Enrollment will begin in 2013, and it aims to have a sample size of 840 subjects in 2 years. The trial is scheduled to complete in 2015.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke, death or cardiovascular events | 30 days
  The participants who suffer from Ischemic stroke, death or cardiovascular events after enrollment or any revascularization procedure of the qualifying lesion in the territory of the symptomatic intracranial artery

SECONDARY OUTCOMES:
Any stroke, or death | beyond 30 days through 6 months
  the number of participants who suffer from any stroke(minor or major, ischemic or bleeding) or death
the number of participants who suffer from restenosis (>50%) related to intracranial stenting | up to 12 months
  the number of participants who suffer from restenosis (>50%) related to intracranial stenting
the changes from baseline in mRS, national institutes of health stroke scale (NIHSS) and Barthel Index | at 7 days, 30 days, 6 months, 12 months, 24 months and 36 months
  the changes from baseline in mRS, national institutes of health stroke scale (NIHSS) and Barthel Index
the number of participants who survives in all patients | beyond 12 months to 36 months
  the number of participants who survives in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ling, MD, Principal Investigator — Xuanwu Hospital, Capital University of Medical Sciences, Beijing, China
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, China

REFERENCES:
- [Result] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Result] Feigin VL. Stroke epidemiology in the developing world. Lancet. 2005 Jun 25-Jul 1;365(9478):2160-1. doi: 10.1016/S0140-6736(05)66755-4. No abstract available. PMID 15978910
- [Result] Zaidat OO, Klucznik R, Alexander MJ, Chaloupka J, Lutsep H, Barnwell S, Mawad M, Lane B, Lynn MJ, Chimowitz M; NIH Multi-center Wingspan Intracranial Stent Registry Study Group. The NIH registry on use of the Wingspan stent for symptomatic 70-99% intracranial arterial stenosis. Neurology. 2008 Apr 22;70(17):1518-24. doi: 10.1212/01.wnl.0000306308.08229.a3. Epub 2008 Jan 30. PMID 18235078
- [Result] Fiorella D, Levy EI, Turk AS, Albuquerque FC, Niemann DB, Aagaard-Kienitz B, Hanel RA, Woo H, Rasmussen PA, Hopkins LN, Masaryk TJ, McDougall CG. US multicenter experience with the wingspan stent system for the treatment of intracranial atheromatous disease: periprocedural results. Stroke. 2007 Mar;38(3):881-7. doi: 10.1161/01.STR.0000257963.65728.e8. Epub 2007 Feb 8. PMID 17290030
- [Result] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Derived] Han Z, Wang T, Li L, Fan J, Wang R, Zheng Y, Yan F, Zhao H, Luo Y, Jiao L. Expression profiles and potential clinical significance of circular RNAs in peripheral neutrophils of patients with intracranial atherosclerotic stenosis. Brain Circ. 2025 Jul 3;11(3):200-211. doi: 10.4103/bc.bc_16_24. eCollection 2025 Jul-Sep. PMID 40842453
- [Derived] Zhao F, Wang T, Luo J, Gao H, Zheng Y, Wang R, Fan J, Zhao H, Han Z, Luo Y, Jiao L. Endothelial Glycocalyx in Cerebral Infarction After Endovascular Treatment in Patients With Intracranial Artery Stenosis. CNS Neurosci Ther. 2025 Aug;31(8):e70545. doi: 10.1111/cns.70545. PMID 40808328